CLINICAL TRIAL: NCT01474785
Title: RYGB Improves Metabolism by Interrupting the Gastric Adipose Tissue Axis
Brief Title: RYGB and the Gastric Adipose Axis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Naji Abumrad, Professor of Surgery, Chairman Department of Surgery, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: #111237; R01DK091748 (NIH)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Nashville, Tennessee
MeSH Terms: conditions — Obesity | interventions — Ghrelin; Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RYGB (Experimental): Roux-en-Y gastric bypass surgery (RYGB) subjects to undergo hyperinsulinemic-euglycemic clamp with human ghrelin infusion pre-operatively and post-operatively.
  Interventions: Drug: human ghrelin; Procedure: Hyperinsulinemic/Euglycemic Clamp
- VSG (Experimental): Vertical sleeve gastrectomy (VSG) subjects to undergo hyperinsulinemic-euglycemic clamp pre-operatively and post-operatively.
  Interventions: Procedure: Hyperinsulinemic/Euglycemic Clamp
- Low Calorie Diet (Experimental): Subjects will receive very low calorie diet prescribed for RYGB patients and undergo hyperinsulinemic-euglycemic before and after diet.
  Interventions: Other: very low calorie diet; Procedure: Hyperinsulinemic/Euglycemic Clamp

INTERVENTIONS:
Drug: human ghrelin — 0.5-1 pmol/kg.min of human ghrelin administered by IV two times
  Arms: RYGB
Other: very low calorie diet — standard very low calorie diet that is prescribed for all RYGB patients after their operation
  Arms: Low Calorie Diet
Procedure: Hyperinsulinemic/Euglycemic Clamp — Insulin and glucose infusions to measure glucose kinetics.

SUMMARY:
The purpose of this study is to determine if interruption in gastric-adipose tissue axis signaling contributes to early improvements in oxidative stress, insulin sensitivity, and inflammation, and to determine if interruption of the stomach in RYGB results in reduction of plasma acylated ghrelin (AG) and in an altered acylated ghrelin:unacylated ghrelin (AG:UAG) ratio which may contribute to decreased oxidative stress and improved insulin sensitivity.

ELIGIBILITY:
PROTOCOL I

Inclusion Criteria:

* Age 18-65 years
* BMI ≥ 35 kg/m^2
* Scheduled for bariatric surgery
* Considering bariatric surgery
* Waiting for insurance approval for bariatric surgery
* Currently not considering bariatric surgery, but otherwise eligible
* Enrollment in medical weight loss program

Exclusion Criteria:

* Smoking >7 cigarettes per day
* Precious malabsorptive or restrictive intestinal surgery
* Pregnant or breastfeeding
* Recent history of neoplasia (5<years ago)
* Malabsorptive syndromes
* Inflammatory intestinal disease
* Established organ disfunction
* Allergy to acetaminophen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
change in glucose disposal rate | baseline and 1 week
  Glucose disposal rate is a sensitive laboratory procedure for determining how your body uses sugar (called insulin sensitivity).

CONTACTS AND LOCATIONS:
Overall Officials: Naji Abumrad, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Flynn CR, Tamboli RA, Antoun J, Sidani RM, Williams B, Spann MD, English WJ, Welch EB, Sundaresan S, Abumrad NN. Caloric Restriction and Weight Loss Are Primary Factors in the Early Tissue-Specific Metabolic Changes After Bariatric Surgery. Diabetes Care. 2022 Aug 1;45(8):1914-1916. doi: 10.2337/dc22-0069. PMID 35724307